CLINICAL TRIAL: NCT07366489
Title: Efficacy and Safety of the RDI Mode in Endoscopic Submucosal Dissection: a Multicenter, Randomized Controlled Study
Brief Title: Efficacy and Safety of the RDI Mode in Endoscopic Submucosal Dissection
Acronym: RM-ESD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Guangdong Second Provincial General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-728
Record Dates: First submitted 2025-12-26; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Endoscopic Submucosal Dissection (ESD)
Keywords: ESD; RDI; early cancer; polyp
MeSH Terms: conditions — Neoplasms; Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDI group (Experimental): Throughout the entire ESD dissection, the RDI mode is used continuously for submucosal dissection (while white-light endoscopy may be employed for observation and marking).
  Interventions: Other: RDI
- WLE group (No Intervention): The WLE group completes the entire ESD procedure using only WLE, without switching to RDI.

INTERVENTIONS:
Other: RDI — Throughout the entire ESD dissection, the RDI mode is used continuously for submucosal dissection (while white-light endoscopy may be employed for observation and marking).
  Arms: RDI group

SUMMARY:
Conventional white-light endoscopy (WLE) is hampered by insufficient contrast when attempting to identify deep vessels and active bleeding sites; visibility drops further when blood pools or spurts obscure the field, resulting in significantly lower hemostatic efficiency. Red dichromatic imaging (RDI), a novel image-enhanced endoscopic modality, has recently been shown to improve the visualization of deep-lying vessels and bleeding points, shorten hemostasis time and potentially increase overall procedural efficiency.

Although retrospective series have suggested that RDI may facilitate intra-operative bleeding control and better delineation of the submucosal plane during endoscopic submucosal dissection (ESD), high-level evidence from multicenter, randomized, controlled trials (RCTs) is lacking. No study has yet demonstrated superiority over WLE with respect to critical endpoints such as en-bloc resection rate, procedure time, complication rate and operator mental workload.

The investigators therefore designed a multicenter RCT to systematically compare the efficacy and safety of full-procedural RDI with conventional WLE during ESD.

The primary outcome parameter is the mean resection speed (mm²/min) achieved with RDI versus conventional white-light endoscopy during ESD.

The secondary outcome parameters are: complete resection (R0) rate, en-bloc resection rate, resection margin, number of intra-procedural bleeding episodes, intra-procedural blood loss, intra-procedural hemostasis time, other intra-procedural adverse events, and post-procedural adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.

  * Early gastric cancer or precancerous lesions, early esophageal cancer or precancerous lesions, or early colorectal cancer/polyps that meet ESD indications.

    * ESD procedure to be performed at a participating center.

      * Lesion diameter 20-60 mm. ⑤ Written informed consent provided voluntarily.

Exclusion Criteria:

① Foreigners.

② Severe coagulopathy (platelet count <50×10⁹/L or INR >1.5), significant cardiopulmonary disease, or any other contraindication to endoscopic therapy.

③ Imaging evidence of distant metastasis or lymph-node metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
mean resection speed (mm²/min) achieved with RDI versus conventional WLE during ESD | Periprocedural
  The resection speed is calculated as the area on the specimen-fixation board divided by the time elapsed from the first mucosal incision to complete dissection of the lesion.

SECONDARY OUTCOMES:
complete resection (R0) rate | Periprocedural
  complete resection (R0) rate
en-bloc resection rate | Periprocedural
  en-bloc resection rate
resection margin | Periprocedural
  vertical and horizontal resection margin
number of intra-procedural bleeding episodes | Periprocedural
  number of intra-procedural bleeding episodes
intra-procedural blood loss | Periprocedural
  intra-procedural blood loss
intra-procedural hemostasis time | Periprocedural
  intra-procedural hemostasis time
other intra-procedural adverse events | Periprocedural
  perforation, infection, and other adverse eventes
post-procedural adverse events | From enrollment to 30 days after the procedure.
  perforation, infection, delayed gastrointestinal bleeding, and other adverse events,

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT07366489/Prot_000.pdf
  • Informed Consent Form (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT07366489/ICF_001.pdf